CLINICAL TRIAL: NCT05521373
Title: Ultrasound-guided Versus Combined Ultrasound and Fluoroscopy-guided Cervical Selective Nerve Root Block for Lower Cervical Radiculopathy: Non-inferiority Randomized Controlled Study
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Nevert Adel, assist. prof. of anesthesia and pain management, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD.22.03.627
Record Dates: First submitted 2022-08-13; First posted 2022-08-30 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Cervical Pain
MeSH Terms: conditions — Neck Pain | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound cervical selective nerve root block (Active Comparator): A (7-12) MHz linear transducer will be applied to the symptomatic side of the neck in the transverse plane. The targeted nerve root of each patient will be identified by moving the transducer cranially from the C7 transverse process as a reference point.
  After the targeted nerve root identified, a needle will be gently introduced toward the dorsal aspect of the nerve root under real-time US guidance with an in-plane approach. The needle tip will be placed between the nerve root and posterior tubercle outside of the intervertebral foramen and the vessels will be around the nerve root with color Doppler. On confirmation of the absence of abnormal findings and careful aspiration, 3 cc of the treatment drug composed of dexamethasone (10 mg) and 0.2% lidocaine, will be injected under real-time US guidance
  Interventions: Device: ultrasound cervical selective nerve root block
- ultrasound and fluoroscopy-guided cervical selective nerve root block (Active Comparator): The targeted transverse process was identified by slowly moving the probe in all directions with the 7th cervical spine transverse process as the reference point. a spinal needle 22 G was inserted. First, 1 ml of the contrast media was injected. The antero-posterior images were obtained to confirm the distribution or spread pattern of the injected contrast media with C-arm fluoroscopy. The following steps were initiated after confirming for proper shadowed contrast of the nerve root and absence of intravascular injection of the contrast media. Three cc of the treatment drug, composed of dexamethasone (10 mg) and 0.5 % lidocaine will be injected after confirming the absence of abnormal findings.
  Interventions: Device: ultrasound and fluoroscopy-guided cervical selective nerve root block

INTERVENTIONS:
Device: ultrasound cervical selective nerve root block — A (7-12) MHz linear transducer will be applied to the symptomatic side of the neck in the transverse plane. The targeted nerve root of each patient will be identified by moving the transducer cranially from the C7 transverse process as a reference point.
  After the targeted nerve root identified, a needle will be gently introduced toward the dorsal aspect of the nerve root under real-time US guidance with an in-plane approach. The needle tip will be placed between the nerve root and posterior tubercle outside of the intervertebral foramen and the vessels will be around the nerve root with color Doppler. On confirmation of the absence of abnormal findings and careful aspiration, 3 cc of the treatment drug composed of dexamethasone (10 mg) and 0.2% lidocaine, will be injected under real-time US guidance
  Arms: ultrasound cervical selective nerve root block
Device: ultrasound and fluoroscopy-guided cervical selective nerve root block — The targeted transverse process was identified by slowly moving the probe in all directions with the 7th cervical spine transverse process as the reference point. a spinal needle 22 G was inserted. First, 1 ml of the contrast media was injected. The antero-posterior images were obtained to confirm the distribution or spread pattern of the injected contrast media with C-arm fluoroscopy. The following steps were initiated after confirming for proper shadowed contrast of the nerve root and absence of intravascular injection of the contrast media. Three cc of the treatment drug, composed of dexamethasone (10 mg) and 0.5 % lidocaine will be injected after confirming the absence of abnormal findings.
  Arms: ultrasound and fluoroscopy-guided cervical selective nerve root block

SUMMARY:
Cervical radiculopathy is a pain and/or sensorimotor deficit syndrome that is defined as being caused by compression of a cervical nerve root .The compression can occur as a result of disc herniation, spondylosis, instability, trauma, or rarely, tumors. Patient presentations can range from complaints of pain, numbness, and/or tingling in the upper extremity to electrical type pains or even weakness. The clinical overlap between cervical radiculopathy and peripheral nerve entrapment syndromes and their nearly ubiquitous nature makes understanding of and identification of these entities mandatory for all practitioners The cervical spinal nerves exit the spinal cord and are oriented obliquely toward their respective neural foramen .The neural foramen is made up of the facet joint posteriorly and the intervertebral disc anteriorly. The superior and inferior borders are comprised of the pedicles of the vertebral bodies above and below, respectively. The foramina are largest in the upper cervical spine and gradually narrow distally, with the C7/T1 foramina being the narrowest. The most common causes of nerve root compression are spondylosis of the facet joint and herniation of the intervertebral disc.Hypermobility of the facet joint leads to ligamentous hypertrophy as well as bony hypertrophy. An increase in the size of the superior articulating process from the distal vertebra causes compression of the nerve. Intervertebral disc herniations can also cause nerve root compression from the anterior aspect of the foramen. Disc herniations can either be acute or chronic.

Imaging modalities and electrophysiologic testing (EMG & NCV) play an important role in the diagnosis and localization of cervical radiculopathy. The first test that is typically done is plain x-ray. Computed tomography is the most sensitive test for examination of the bony structures of the spine.

Initial strategies in the treatment of cervical radiculopathy are typically Conservative therapies including multiple pharmacologic agents, immobilization, physical therapy, manipulation, traction, and TENS .

Traditionally, cervical spine injection performed under fluoroscopy or computed tomography guidance. However, these imaging tools are not able to visualize small vessels, and incidences such as brainstem or spinal cord infarction may occur. These complications are believed to be caused by inadvertent injection of therapeutic agents into the vertebral or radicular arteries. Therefore, accidental puncture of vessels must be prevented when performing neck injection procedures.

Recently, high-resolution musculoskeletal ultrasound (US) can be used to identify the target root and the nearby vessels. The advantage of using US as a guidance tool is that it does not expose patients or medical personnel to radiation such as fluoroscopy or computed tomography guidance. Ultrasound allows good visualization of the soft tissue such as abnormal blood vessels in the foramen and around the nerve root, which further enables accurate needle placement and avoids the risk of intravascular injections. In addition, US-guided procedures have a shorter duration compared to those guided by fluoroscopy and do not result in contrast medium-related allergic reactions . As a result, US-guided cervical nerve root block (US-CRB) is a safe alternative treatment technique that can be used in the treatment of upper extremity radicular pain.

DETAILED DESCRIPTION:
This study will be conducted to evaluate immediate and long-term effectiveness, functional improvements, and safety of ultrasound (US)-guided selective cervical nerve root block compared with fluoroscopy-guided selective nerve root block.

Technique of ultrasound guided cervical selective nerve root block:

Basic monitoring with non-invasive arterial blood pressure, electrocardiogram and pulse oximetry will be applied before the procedure, an intravenous catheter (20 G) will be inserted in a peripheral line for crystalloid infusion. Patients will be positioned in the oblique supine decubitus position with head externally rotated at 30° to 40° away from the targeted area, the frontal cervical spine area from the clavicle to mandible was adequately disinfected with Betadine and an aseptic dressing was applied. The sternocleidomastoid muscle was first palpated from the posterior side to palpate the transverse process of the cervical spine.

A (7-12) MHz linear transducer of a US machine will be applied to the symptomatic side of the neck in the transverse plane. Initially, the cervical nerve roots will be identified on US by the shape of the transverse process. Unlike the transverse processes of the 3rd to 6th cervical spines, the transverse process of the 7th cervical spine has a rudimentary anterior tubercle and a prominent posterior tubercle. The C6 transverse process characterized by its sharp anterior tubercle. The C5 transverse process identified by the "two-humped camel" sign formed by anterior and posterior tubercles. Within the intertubercular groove of the corresponding transverse process, the nerve root of each cervical spinal level will be observed with hypoechoic texture. The targeted nerve root of each patient will be identified by moving the transducer cranially from the C7 transverse process as a reference point.

The optimal image of the nerve root, location of the radicular artery and surrounding vessels near the border of the nerve root were obtained through probe manipulation in the power and color Doppler modes After the targeted nerve root identified, a 60-mm, 23-G needle will be gently introduced toward the dorsal aspect of the nerve root under real-time US guidance. The needle will be inserted just lateral to the transducer and advanced, from postero-lateral to antero-medial, with an in-plane approach. The needle tip will be placed between the nerve root and posterior tubercle outside of the intervertebral foramen and approached close to the epineurium with care to avoid inadvertent injection to the vessel through locating the vessels around the nerve root with color Doppler. Then, 1 ml of 1% lidocaine will be injected, following which the patient monitored for the onset of clinical manifestations such as mid-neck and contralateral arm pain, metallic taste, dizziness, tachycardia, full-body paraesthesia, auditory changes, slurred speech, and motor ataxia for 1 to 2 minutes. On confirmation of the absence of abnormal findings and careful aspiration, 3 cc of the treatment drug composed of dexamethasone (10 mg) and 0.5% lidocaine, will be injected under real-time US guidance

Technique of combined ultrasound and fluoroscopy guided selective nerve root block:

With the patient's head externally rotated 30 to 40 degrees away from the targeted area in a supine position, the frontal cervical spine area from the clavicle to mandible was adequately disinfected with Betadine and an aseptic dressing was applied. The sternocleidomastoid muscle was first palpated from the posterior side to palpate the transverse process of the cervical spine. A probe was placed and a transverse scan image of the transverse process was obtained after locating the transverse process. The location of the 7th transverse process was confirmed by visualization of the adjacent transverse processes sonographically from the superior to inferior direction. Unlike the transverse processes of the 3rd to 6th cervical spines, the transverse process of the 7th cervical spine has a rudimentary anterior tubercle and a prominent posterior tubercle, a unique characteristic used to identify and differentiate the 7th transverse process.

The targeted transverse process was identified by slowly moving the probe in all directions with the 7th cervical spine transverse process as the reference point. The optimal image of the nerve root, the location of the radicular artery, and the surrounding vessels near the border of the nerve root were obtained through the probe manipulation. Next, a spine needle 22 G was inserted from the posterior to anterior direction, toward the nerve root and parallel to the probe. The needle end was placed on the dorsal side of the nerve by cautiously avoiding damage to the possible deep cervical artery near the insertion site and locating the area free of the radicular artery. First, 1 ml of the contrast media was injected. The antero-posterior images were obtained to confirm the distribution or spread pattern of the injected contrast media with C-arm fluoroscopy. The following steps were initiated after confirming for proper shadowed contrast of the nerve root and absence of intravascular injection of the contrast media. One millilitre of 1 % lidocaine was injected and monitored for the onset of clinical manifestations such as mid-neck and contralateral arm pain, metallic taste, dizziness, tachycardia, full body paraesthesia, auditory changes, slurred speech, and motor ataxia for 1-2 min. Three cc of the treatment drug, composed of dexamethasone (10 mg) and 0.5 % lidocaine will be injected after confirming the absence of abnormal findings. The procedure will be completed after obtaining the images of the wash out spot

ELIGIBILITY:
Inclusion Criteria:

* • Patients between 18-80 years old

  * Both sexes.
  * Single level cervical radiculopathy C6 or C7.
  * Cervical radicular pain was diagnosed on the basis of clinical profiles, medical examinations
  * Radiologic finding via cervical computed tomography or magnetic resonance imaging was consistent with the clinical diagnosis.
  * Patients presenting with acute and sever symptoms with verbal numeric scale (VNS) at least 5 points for at least 3 months prior to study entry (day 0)
  * Pain relief not achieved with conservative treatments administered for at least 4 weeks, including analgesic use (nonsteroidal anti-inflammatory drugs (NSAIDs) or opioids) and physical therapy.

Exclusion Criteria:

* • Patients younger than 18 years or older than 80 years.

  * Patient refusal.
  * Pregnant or lactating women.
  * Psychiatric disorders affecting co-operation of the patient.
  * Bleeding or coagulation disorders
  * Local skin infection or current other problem in the affected extremity.
  * Prior allergic reaction to any of the study medications; contrast media, steroid or local anaesthetic.
  * Laboratory result suggestive of systemic inflammatory disease or rheumatoid disorder.
  * Cervical radiculopathy at multiple levels.
  * Cervical myelopathy.
  * Patient presenting with motor power less than Medical Research Council MRC grade 4.
  * Injections within prior 3 months.
  * Recent cervical spinal surgery.
  * Previous chronic opioid use.
  * Any condition that could interfere with the interpretation of the outcome assessments.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Numerical rating scale | immediately before Cervical Selective Nerve Root Block
  0=no pain , 10=sever pain
Numerical rating scale | after 2 weeks from Cervical Selective Nerve Root Block
  0=no pain , 10=sever pain
Numerical rating scale | after 1 month from Cervical Selective Nerve Root Block
  0=no pain , 10=sever pain
Numerical rating scale | after 2 months from Cervical Selective Nerve Root Block
  0=no pain , 10=sever pain
Numerical rating scale | after 3 months from Cervical Selective Nerve Root Block
  0=no pain , 10=sever pain
neck disability index questionnaire | immediately before Cervical Selective Nerve Root Block
  it is a questionnaire composed of 10 items: pain, Personal Care, Lifting, Reading, Headaches, Concentration, Work, Driving, Sleeping, Recreation. each item ranges from 0= do not affect to 5= worst affect and the total score of the 10 items will be summed. if the total score will be 4 or lower, no disability; 5 to 14, mild disability; 15 to 24, moderate disability; 25 to 34, severe disability; 35 or over, complete disability.
neck disability index questionnaire | after 1 month from Cervical Selective Nerve Root Block
  it is a questionnaire composed of 10 items: pain, Personal Care, Lifting, Reading, Headaches, Concentration, Work, Driving, Sleeping, Recreation. each item ranges from 0= do not affect to 5= worst affect and the total score of the 10 items will be summed. if the total score will be 4 or lower, no disability; 5 to 14, mild disability; 15 to 24, moderate disability; 25 to 34, severe disability; 35 or over, complete disability.
neck disability index questionnaire | after 2 months from Cervical Selective Nerve Root Block
  it is a questionnaire composed of 10 items: pain, Personal Care, Lifting, Reading, Headaches, Concentration, Work, Driving, Sleeping, Recreation. each item ranges from 0= do not affect to 5= worst affect and the total score of the 10 items will be summed. if the total score will be 4 or lower, no disability; 5 to 14, mild disability; 15 to 24, moderate disability; 25 to 34, severe disability; 35 or over, complete disability.
neck disability index questionnaire | after 3 months from Cervical Selective Nerve Root Block
  it is a questionnaire composed of 10 items: pain, Personal Care, Lifting, Reading, Headaches, Concentration, Work, Driving, Sleeping, Recreation. each item ranges from 0= do not affect to 5= worst affect and the total score of the 10 items will be summed. if the total score will be 4 or lower, no disability; 5 to 14, mild disability; 15 to 24, moderate disability; 25 to 34, severe disability; 35 or over, complete disability.

SECONDARY OUTCOMES:
time of the procedure by minutes | during the injection procedure
  starting from putting the ultrasound probe until withdraw the needle after injection
patient satisfaction from 0 to 10 | after two months from Cervical Selective Nerve Root Block
  0 = not satisfied , 10 = maximum satisfied
complication | during the performance of the procedure
  any complication during the procedure as intravascular injection, hypotension, bradycardia

CONTACTS AND LOCATIONS:
Locations (1):
- Yahya Wahba, Al Mansurah, Egypt